CLINICAL TRIAL: NCT04013178
Title: Eccentric Exercise and Electromyostimulation to Improve Muscle Strength and Muscle Mass After Radiation Therapy for Head and Neck Cancer
Brief Title: Exercise After Radiation for Head & Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Guillaume Millet, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-16-0744
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accentuated eccentric loading + electromyostimulation (Experimental): This group will undertake a supervised 12-week intervention involving accentuated eccentric loading and electromyostimulation of the knee extensors, dynamic resistance training of lower limb antagonist and synergist muscles and upper limb dynamic resistance training.
  Interventions: Behavioral: Accentuated eccentric loading + electromyostimulation
- Traditional resistance training (Active Comparator): This group with undertake a supervised 12-week intervention involving volume matched dynamic resistance training of the knee extensors, and dynamic resistance training of lower limb antagonist and synergist muscles and upper limb dynamic resistance training.
  Interventions: Behavioral: Conventional resistance training

INTERVENTIONS:
Behavioral: Accentuated eccentric loading + electromyostimulation — An innovative training intervention to optimize muscle strength and muscle mass
  Arms: Accentuated eccentric loading + electromyostimulation
Behavioral: Conventional resistance training — A conventional approach to resistance training
  Arms: Traditional resistance training

SUMMARY:
People who receive radiation therapy for head and neck cancer (HNC) can experience side-effects which include a significant loss in body mass and a loss of muscle mass (cancer cachexia). Some research has shown success in the use of generic (dynamic) resistance training interventions for patients affected by head and neck cancer. However, this approach could be optimized with the use of novel training methods.The primary aim of this research is to investigate the effect of conventional resistance training vs. an experimental intervention (electromyostimulation combined with accentuated eccentric loading) on muscle strength and muscle mass after radiation for HNC.

DETAILED DESCRIPTION:
Background and Rationale

Patients who receive radiation therapy for head and neck cancer treatment are susceptible to side-effects such as a significant loss in body mass and a loss of muscle mass (cancer cachexia) compared to pre-treatment. In addition, radiation therapy treatment may cause cancer-related fatigue and a reduction in overall physical function and health-related quality of life. Some research has shown success in the use of generic (dynamic exercise) resistance training interventions when applied for head and neck cancer survivors. Typically, when the correct training principals are adhered to in healthy populations (i.e. progressive overload, specificity, variation, rest/recovery), muscle strength and muscle mass are effectively enhanced. However, these training variables may be less effective in eliciting positive outcomes in clinical populations in that they are less effective in increasing muscle mass and muscle strength. Exercise is beneficial for people affected by all cancer types, but resistance training may be particularly beneficial for people who have completed radiation therapy treatment for head and neck cancer. Alternative modalities may provide superior improvements in muscle strength and muscle mass. Therefore, further research is warranted to investigate optimized resistance training prescription in head and neck cancer patients.

Research Question & Objectives

The primary aim of this research is to investigate the effect of conventional resistance training vs. an experimental intervention (electromyostimulation combined with accentuated eccentric loading) on muscle strength and muscle mass after radiation for HNC.

Methods

Head and neck cancer survivors who have completed radiation therapy ≥ 1 month and ≤ 1 year from enrollment will be randomly allocated to one of two treatment arms: conventional (active control) and accentuated eccentric loading + electromyostimulation. Participants will be assessed before and after the intervention for patient-reported outcomes, neuromuscular function and fatigability in response to whole-body exercise.

ELIGIBILITY:
Inclusion Criteria:

* a verified clinical diagnosis of head and neck cancer (stage I-IV) with the primary tumor in the oral cavity, pharynx, larynx, paranasal sinuses, or salivary glands.
* received radiation therapy ± concomitant chemotherapy
* able to walk without assistance
* received Canadian Society for Exercise Physiology-Certified Exercise Physiologist (CSEP-CEP) approval via The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and/or physician approval
* willing/able to travel to the University of Calgary (Calgary, AB).

Exclusion Criteria:

* comorbidities that could confound the ability to participate in laboratory tests (e.g. other malignancies, neuromuscular, musculoskeletal or vascular conditions affecting the lower extremities, such as radiculopathy or myopathy, (where the research team were consulted for individual cases)
* presence of a percutaneous endoscopic gastrostomy
* unable to follow verbal instructions in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2020-06-26 (Estimated)

PRIMARY OUTCOMES:
Maximal Isometric Force in the Knee Extensors | Baseline and after the 12-week intervention
  A change in maximal isometric force in the knee extensors measured before, during and after an intermittent cycling test.
Assessment of change in Muscle Cross-Sectional Area | Baseline and after the 12-week intervention
  ultrasound measurement of the vastus lateralis and rectus femoris

SECONDARY OUTCOMES:
Assessment of change in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Scale | Baseline to after the 12-week intervention, at 6 month and 12 month follow up
  Self-report questionnaire for the assessment of cancer-related fatigue. This scale is between a possible raw score of 0 - 52, where the higher the number, the better the outcome.
Assessment of change in the Functional Assessment of Chronic Therapy - Head and Neck (FACT-H&N) Scale | Baseline to after the 12-week intervention, at 6 month and 12 month follow up
  Self-report questionnaire for the assessment of quality of life. This scale is between a possible 0 - 144 points, where the higher the number the better the outcome. There are 5 individual sub scales that measure physical-, social-, emotional-, and functional well-being as well as head and neck specific concerns.
Voluntary Activation | Baseline and after the 12-week intervention
  A reduction voluntary activation (using femoral nerve stimulation) measured before, during and after an intermittent cycling test
Potentiated Twitch Force | Baseline and after the 12-week intervention
  A reduction in potentiated quadriceps twitch force measured before, before, during and after an intermittent cycling test.
Muscle Compound Action Potential (M-Wave) Peak-to Peak Amplitude | Baseline and after the 12-week intervention
  evoked from supra-maximal stimulation of the femoral nerve and measured before, during and after an intermittent cycling test
Voluntary Electromyography (EMG) | Baseline and after the 12-week intervention
  Root mean square of the EMG signal during an MVC, measured before, during and after an intermittent cycling test.
Time to volitional exhaustion | Baseline and after the 12-week intervention
  Time to task failure during an intermittent cycling test
Body mass (kg) | Baseline and after the 12-week intervention
Estimated body fat % | Baseline and after the 12-week intervention
  Estimated using skin folds
Body mass index | Baseline and after the 12-week intervention
  Body mass / (height * height)

CONTACTS AND LOCATIONS:
Overall Officials: Gui Millet, PhD, Principal Investigator — University of Calgary
Locations (1):
- Faculty of Kinesiology, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No